CLINICAL TRIAL: NCT07082179
Title: The Efficacy and Safety of Iparomlimab and Tuvonralimab Combined With Paclitaxel Polymer Micelles and Platinum (Cisplatin/Carboplatin) in the Treatment of Stage III Unresectable Non-small Cell Lung Cancer
Brief Title: A Prospective Phase II Clinical Study of Immunotherapy Combined With Chemotherapy for Stage III Unresectable Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Meiqi Shi, Chief Physician, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jiangsu Cancer Hospital
Record Dates: First submitted 2025-07-07; First posted 2025-07-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: NSCLC
Keywords: Iparomlimab and Tuvonralimab,Chemotherapy, unresectable non-small cell lung cancer
MeSH Terms: interventions — Platinum; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Iparomlimab and Tuvonralimab combined with paclitaxel polymer micelles and Platinum (cisplatin/carboplatin)
  Interventions: Drug: Iparomlimab and Tuvonralimab combined with paclitaxel polymer micelles and Platinum (cisplatin/carboplatin)

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab combined with paclitaxel polymer micelles and Platinum (cisplatin/carboplatin) — The induction therapy regimen is as follows: Apalotamab: 5 mg/kg, every 3 weeks (q3w), administered via intravenous infusion. Paclitaxel polymer micelles in combination with platinum: In cycle 1, paclitaxel polymer micelles 230 mg/m² administered via intravenous infusion over ≥3 hours, with the option to escalate the dose in cycle 2 according to the instructions for use, followed by cisplatin 70 mg/m² or carboplatin AUC 5 mg/mL/min. The local treatment regimen involves re-evaluation by a multidisciplinary team (MDT), surgery, or radical radiotherapy or single fractionated segmental radiotherapy (two radiotherapy regimens for the investigator to choose from). The consolidation therapy regimen consists of apalotamab consolidation for 1 year or up to a maximum of 17 cycles, with the decision to combine with chemotherapy left to the discretion of the treating physician on an individual basis.

SUMMARY:
This study is a prospective, multicenter, open-label, single-arm Phase II clinical trial. The study recruits patients with stage III unresectable non-small cell lung cancer according to the 8th edition of the AJCC/UICC staging system. It aims to observe and evaluate the efficacy and safety of anti-PD-1/CTLA-4 antibody in combination with paclitaxel polymer micelles and platinum-based therapy for stage III unresectable non-small cell lung cancer.

DETAILED DESCRIPTION:
This study includes a screening period (the maximum time interval from screening to the start of treatment ≤21 days), a treatment period (including the induction therapy phase, local therapy phase [surgery or radiotherapy], and consolidation therapy phase), and a follow-up period (including safety follow-up and survival follow-up). The primary endpoint is the objective response rate after induction therapy. Secondary endpoints include the pathological complete response rate in operable patients, major pathological response rate, surgical conversion rate, R0 resection rate, and 18-month event-free survival rate, among others.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males or females aged 18 to 75 years.
* 2. Histologically or cytologically confirmed squamous or non-squamous (EGFR/ALK/ROS1 negative) non-small cell lung cancer.
* 3. No prior local treatment (surgery or radiotherapy) or any systemic anti-tumor treatment for the tumor, including cytotoxic therapy, targeted therapy (including tyrosine kinase inhibitors or monoclonal antibodies), cell therapy, immunotherapy, traditional Chinese medicine treatment, or any other investigational drug treatment.
* 4. Patients with unresectable stage III disease (according to the 8th edition AJCC TNM staging for non-small cell lung cancer, T1-2N2-3M0, T3N1-3M0, T4N0-3M0) after multidisciplinary team (MDT) assessment.
* 5. At least one measurable lesion according to RECIST v1.1 criteria, as shown by chest enhanced CT or PET/CT.
* 6. ECOG performance status: 0 or 1.
* 7. The patient is able to tolerate induction therapy and surgery. Radical surgical resection and systematic lymph node dissection are recommended, provided that surgical margins can be ensured and the patient's general condition is taken into account.
* 8. Expected survival of ≥12 months.
* 9. Major organ and marrow function meet the following requirements:
* Hematologic tests (no transfusions or blood products, no use of G-CSF or other hematopoietic growth factors within 14 days):

  1. Hematologic indices: Absolute neutrophil count ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥90 g/L.
  2. Liver and kidney function indices: Total bilirubin ≤1.5×ULN, ALT/AST ≤2.5×ULN; creatinine ≤1.5×ULN, or creatinine clearance ≥60 mL/min; urine routine test with proteinuria less than 2+. If the patient has proteinuria ≥2+ at baseline, a 24-hour urine collection should be performed to demonstrate that the 24-hour urine protein quantification is ≤1 g.
  3. Coagulation function indices: INR ≤1.5; activated partial thromboplastin time (APTT) ≤1.5×ULN.
  4. Endocrine system: Thyroid-stimulating hormone (TSH) within normal limits. Note: If TSH is not within the normal range at baseline, but T3 and free T4 are within the normal range, the subject is still eligible.
* Cardiopulmonary function meets the following requirements:

  1. Pulmonary function indices: FEV1.0 > 1.0 L or FEV% > 50%.
  2. Cardiac function indices: Electrocardiogram (ECG) QTc interval > 480 msec (QTc interval calculated using the Fridericia formula).
* 10. Women of childbearing potential must have used reliable contraception or have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and agree to use appropriate contraception during the trial and for 8 weeks after the last administration of the investigational drug. For men, they must agree to use appropriate contraception during the trial and for 8 weeks after the last administration of the investigational drug or have undergone surgical sterilization.
* 11. The subject voluntarily agrees to participate in this study, signs the informed consent form, is compliant, and is willing to cooperate with follow-up.

Exclusion Criteria:

* 1. Presence of contraindications to immunotherapy (including long-term use of corticosteroids, history of radiation pneumonitis, etc.).
* 2. History of severe allergy to paclitaxel, docetaxel, platinum agents, or their prophylactic medications.
* 3. Any unstable systemic disease, including active infection, uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg despite optimal medical therapy), unstable angina, angina attack within the past 3 months, liver disease requiring medication, kidney disease, or metabolic disease.
* 4. Received live vaccine within 28 days prior to treatment.
* 5. Previously received radiotherapy, chemotherapy, targeted therapy, or immunotherapy.
* 6. Active autoimmune disease (such as vitiligo, psoriasis, hypothyroidism requiring hormone replacement therapy, etc.).
* 7. Patients with active hepatitis B or C, HIV patients, active tuberculosis, etc.
* 8. Active infection requiring antimicrobial treatment (e.g., requiring antibiotics, antiviral agents, antifungal agents).
* 9. Known history of allogeneic organ transplantation and known history of hematopoietic stem cell transplantation.
* 10. Patients with interstitial lung disease or a history of interstitial pneumonia.
* 11. History of drug abuse or mental disorders that cannot be controlled.
* 12. Previous or concurrent other untreated malignancies, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, and superficial bladder cancer.
* 13. Pregnant or breastfeeding women; patients of childbearing potential who are unwilling or unable to take effective contraceptive measures.
* 14. Other situations that the investigator judges may affect the conduct of the clinical study or the determination of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate ,ORR | Approximately four months

SECONDARY OUTCOMES:
Pathological complete remission rate, pCR | Approximately four months
Major pathological response rate , MPR | Approximately four months
Surgical conversion rate, SCR | Approximately four months
R0 resection rate | Approximately four months
18-month event-free survival rate | 18-month
Event Free Survival，EFS | up to 5 years after treatment discontinuation
Overall survival ,OS | up to 5 years after treatment discontinuation
Safety | From ICF through 100 days after the last dose of study treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
PD-L1 expression | Within 3 years
Tumor mutation burden (TMB) | Within 3 years
Next-generation sequencing (NGS), and chemotherapy drug sensitivity analysis | Within 3 years
  First, use NGS to identify the molecular characteristics of the tumor, and then infer or experimentally verify its sensitivity to specific chemotherapeutic drugs based on these characteristics, thereby achieving precision medicine in clinical practice or research.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Cancer Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No